CLINICAL TRIAL: NCT05109819
Title: ESO-SPARE: Esophagus Sparring Radiotherapy for Thoracic and Cervical Metastatic Spinal Cord Compression. A Randomized Phase III Study.
Brief Title: Esophagus-sparing Radiotherapy for Metastatic Spinal Cord Compression.
Acronym: ESO-SPARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Danish Cancer Society (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Anna Mann Nielsen, Principal Investigator, MD, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AA 2112 ESO-SPARE; H-20069184 (Registry Identifier: Regional Committee on Health Research Ethics, Capital Region, Denmark)
Record Dates: First submitted 2021-10-07; First posted 2021-11-05 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Spinal Cord Compression; Radiation Toxicity; Esophagitis; Patient Reported Outcome Measures
Keywords: Metastatic Spinal Cord Compression; Radiation Toxicity; Esophagitis; Patient reported outcome measures; Palliative radiotherapy
MeSH Terms: conditions — Spinal Cord Compression; Radiation Injuries; Esophagitis

STUDY DESIGN:
Intervention Model Description: Patients with metastatic spinal cord compression in the cervical and/or thoracic spine are randomized into two groups. Group A receives standard radiotherapy, group B receives esophagus sparing therapy.
Who Masked: Participant
Masking Description: The outcome of randomization is not reviled to the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: standard radiotherapy treatment (No Intervention): Patients in arm A will receive standard radiotherapy treatment for metastatic spinal cord compression.
- Arm B: esophagus sparring radiotherapy treatment (Experimental): Patients in arm B will receive esophagus sparring radiotherapy treatment.
  Interventions: Radiation: Esophagus sparring radiotherapy treatment

INTERVENTIONS:
Radiation: Esophagus sparring radiotherapy treatment — A radiotherapy plan for metastatic spinal cord compression is conducted with specific constrains sparring the esophagus.
  Arms: Arm B: esophagus sparring radiotherapy treatment

SUMMARY:
Metastatic spinal cord compression (MSCC) is a serious complication to metastatic cancer and when diagnosed life expectancy is short. Treatment is palliative radiotherapy (RT). Early esophageal toxicity is underreported but can seriously impact quality of life (QoL).

The aim of the ESO-SPARE trial is to investigate if esophagus sparing RT can decrease patient reported esophageal toxicity without compromising ambulatory function or increase other toxicities.

200 patients with MSCC in the thoracic or cervical spine referred for RT will be randomized to either standard or esophagus/pharynx sparing RT. Subsequently participants will be followed with PROM (Patient Reported Outcome Measures) for 9 weeks. PROM-CTCAE questionnaires on upper GI toxicity and pain will be collected daily for 5 weeks and weekly for 4 weeks. Questionnaires evaluating QoL and physical function will be collected weekly for 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histology or cytology proven cancer
* Referred for palliative radiotherapy of the cervical or thoracic vertebra for

  * epidural ingrowth
  * metastatic spinal cord compression
  * metastatic spinal nerve root compression
  * post-operative radiotherapy after decompressive surgery for spinal cord or nerve root compression
* Ability to understand and the willingness to sign a written informed consent document
* Referred for the following dose prescriptions 5 Gy x 5, 5 Gy x 4, 3 Gy x 10, 10 Gy x 1, 8 Gy x 1.
* ≥ 18 years old.

Exclusion Criteria:

- Referred for > 10 fractions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Early patient reported gastro-oesophageal toxicity | Measured within the first 5 weeks after treatment start
  Measured as a peak score using CTCAE Patient Reported Outcome Measures
Ambulatory function | Measured 9 weeks after treatment start
  Preserved ability to walk will be evaluated using the European Quality of Life - 5 Dimensions questionnaire (EQ-5D-5L) mobility dimension. The EQ-5D includes one question for each of the five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5).

SECONDARY OUTCOMES:
Duration of gastro-oesophageal toxicity | Assessed 9 weeks after treatment start
  Measured as the time from an increase in gastro-oesophageal symptom score to a return to baseline
Reirradiation rate - Overall survival (OS) | Assessed 6 months after inclusion of the last patient.
  Defined as fraction of patients getting reirradiation, where the same spine levels are included in the irradiated volume
Patient reported physical function | Assessed Weekly over a period of 9 weeks
  Patient reported physical function will be assessed using answers from the EORTC QLQ-C30 questionnaire. Questions regarding physical function are measured on a four-point scale (1= not at all, 2 = a little, 3 = quite a bit, 4 = very much). All EORTC QLQ-C30 answers will be scored according to the EORTC QLQ-C30 Scoring Manual.
Health related Quality of life (QoL) | Assessed Weekly over a period of 9 weeks
  Health related quality of life measured with EQ-5D-5L European Quality of Life - 5 Dimensions questionnaire (EQ-5D-5L).
  The EQ-5D includes one question for each of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). Health state scores are defined by combining one level from each dimension, ranging from 11111 (full health) to 55555 (worst health).
  A visual analogue scale indicating the respondent's own assessment of their health status from 0-100 is also included (100 = the best health you can imagine and 0 = the worst health you can imagine).
Health related Quality of life (QoL) | Assessed Weekly over a period of 9 weeks
  Health related quality of life assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of life Questionnaire - Cancer (QLQ-C30). The EORTC QLQ-C30 consists of 30 questions assessing quality of life issues using a four-point scale (1= not at all, 2 = a little, 3 = quite a bit, 4 = very much) except from the last two questions which are measured between 1 (Very Poor) to 7 (Excellent). The EORTC QLQ-C30 will be scored according to the EORTC QLQ-C30 Scoring Manual.
Weight | Assessed Weekly over a period of 9 weeks
  Assessed Weekly over a period of 9 weeks
Analgesic consumption | Assessed Weekly over a period of 9 weeks
  Assessed Weekly over a period of 9 weeks
Pain (MSCC site) | Assessed daily for 5 weeks and subsequently weekly for 4 weeks.
  Evaluated by "Numeric Pain Rating Scale (NPRS)"
  The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Pain assessment (MTS site) | Best response during 9 weeks of follow-up
  Assessment will be performed using International Consensus Pain Response Endpoints (ICPRE).
  * A complete pain response is defined as a pain score of 0 out of 10 at the treated site with no concomitant increase in analgesic intake
  * A partial pain response is defined as a pain reduction of 2 or more at the treated site without analgesic increase, or an analgesic reduction of 25% with no increase in pain score or 1 point above baseline.
  * Pain progression is defined as an increase in pain score of 2 or more above baseline with stable analgesic intake or an analgesic increase of 25% with stable pain score.
  * An indeterminate response is any response not captured in the above definitions.
  Analysis of pain reduction will only include patients with NPRS ≥ 1 registered at baseline. We intend to report the best response during follow-up.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Herlev Hospatal, Herlev

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Rabin R, de Charro F. EQ-5D: a measure of health status from the EuroQol Group. Ann Med. 2001 Jul;33(5):337-43. doi: 10.3109/07853890109002087. PMID 11491192

DOCUMENTS (2):
  • Study Protocol (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT05109819/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-29): https://cdn.clinicaltrials.gov/large-docs/19/NCT05109819/SAP_001.pdf